CLINICAL TRIAL: NCT03193645
Title: Observational Prospective Study Describing the Global Patient Care and Follow-up of Prostate Cancer Patients Treated With Degarelix (DUO)
Brief Title: Observational Prospective Study Describing the Global Patient Care and Follow-up of Prostate Cancer Patients Treated With Degarelix
Acronym: DUO
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000235
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Degarelix
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Injection
  Other Names: Firmagon

SUMMARY:
The DUO study's main objective is to evaluate, in the real life, the prevalence of cardiovascular risk in patients with prostate cancer that hormone treatment of androgen suppression by Degarelix was introduced.

This study will also assess, at the initiation of therapy, the prevalence of osteoporosis, metabolic comorbidities, depression, sexual and geriatric patients suffering from prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years or older
* Diagnosed with prostate cancer
* Patient having received an antagonist of GnRH Degarelix prescription.
* Agreeing to and capable of completing in French during the visits all questionnaires on the impact of their illness and treatment.
* Patients having received oral and written study information, agreeing to the use of his anonymized data, and having signed a written Informed Consent Form.

Exclusion Criteria:

* Patient included in an interventional study assessing treatment for prostate cancer.
* Patient presenting hypersensitivity to Degarelix or one of its excipients.
* Patient treated by other hormonotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate gland required.
Study Population: Patients will be enrolled by urologists in private clinics or hospital clinics.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of cardiovascular comorbidity | At inclusion
  Measured by a history of at least one cardiovascular illness (according to ICD-10) and/or at least three cardiovascular risk factors (as defined by Cancer Committee of the French Urology Association)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hopital de la Source (there may be multiple sites in this country), Orléans, France